CLINICAL TRIAL: NCT04337359
Title: Ruxolitinib Managed Access Program (MAP) for Patients Diagnosed With Severe/Very Severe COVID-19 Illness
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Novartis is the Marketing Authorization Holder for Jakavi outside the US. (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424A2001M
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Severe/Very Severe COVID-19 Illness
Keywords: Corona Virus; Pneumonia; Virus; Covid-19; Covid
MeSH Terms: conditions — Pneumonia; Virus Diseases; COVID-19 | interventions — ruxolitinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg. Tablet
  Other Names: Jakavi

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to ruxolitinib for eligible patients diagnosed with severe/very severe COVID-19 illness. The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

The requesting Treating Physician submitted a request for access to drug (often referred to as Compassionate Use) to Novartis which was reviewed and approved by the medical team experienced with the drug and indication.

Please refer to the latest Investigator's Brochure (IB) or approved label for overview of ruxolitinib including: non-clinical and clinical experience, risk and benefits. Novartis will continue to provide any new safety information to the Treating Physician as they emerge.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

Written patient informed consent or assent must be obtained prior to start of treatment.

* Patients aged ≥ 6 years
* Patients clinically diagnosed with SARS-CoV-2 infection, either through positive serum antibodies (IgM or IgG); or by PCR; or by other approved diagnostic methodology. Patients with presumptive diagnosis of COVID-19 (other respiratory causes ruled out and SARS-CoV-2 test pending) may be included.
* Adult and adolescent patients (≥12years), who meet one of the below criteria

  * Respiratory frequency ≥ 30/min
  * Oxygen saturation ≤ 93% on room air (FiO2=0.21)
  * Arterial oxygen partial pressure (PaO2)/ fraction of inspired oxygen (FiO2) <300mmHg(1mmHg=0.133kPa) (corrective formulation should be used for higher altitude regions (over 1000m).

AND

-- Patients with lung imaging showing pulmonary infiltrates (chest X-ray or CT scan)

Pediatric patients (≥6-<12 years) who meet one of the below criteria (where appropriate):

* Shortness of breath
* Oxygen saturation <92% on room air (Fi)2=0.21)
* Labored breathing (e.g. wheezing, flaring of nostrils, three concave sign), cyanosis, intermittent apnea.
* Lethargy or convulsions
* Refusal to eat or difficulty with feeding; signs of dehydration

Exclusion Criteria:

* Patients eligible for this Treatment Plan must not meet any of the following criteria:
* History of hypersensitivity to any drugs or metabolites of similar chemical classes as ruxolitinib
* Presence of severely impaired renal function defined by serum creatinine > 2 mg/dL (>176.8 μmol/L), or have estimated creatinine clearance < 30 ml/min measured or calculated by Cockroft Gault equation or calculated by the updated bedside Schwartz equation.
* Pregnant or nursing (lactating) women.
* Patients who are NOT able to understand and to comply with treatment instructions and requirements unless health care proxy is able to provide consent.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

REFERENCES:
- [Derived] Stanevich OV, Fomina DS, Bakulin IG, Galeev SI, Bakin EA, Belash VA, Kulikov AN, Lebedeva AA, Lioznov DA, Polushin YS, Shlyk IV, Vorobyev EA, Vorobyeva SV, Surovceva TV, Bakulina NV, Lysenko MA, Moiseev IS. Ruxolitinib versus dexamethasone in hospitalized adults with COVID-19: multicenter matched cohort study. BMC Infect Dis. 2021 Dec 22;21(1):1277. doi: 10.1186/s12879-021-06982-z. PMID 34937556
- [Derived] D'Alessio A, Del Poggio P, Bracchi F, Cesana G, Sertori N, Di Mauro D, Fargnoli A, Motta M, Giussani C, Moro P, Vitale G, Giacomini M, Borra G. Low-dose ruxolitinib plus steroid in severe SARS-CoV-2 pneumonia. Leukemia. 2021 Feb;35(2):635-638. doi: 10.1038/s41375-020-01087-z. Epub 2020 Nov 10. No abstract available. PMID 33173161